CLINICAL TRIAL: NCT03368872
Title: Protocol for a Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Impact of a Daily Dose of an Astaxanthin Formulation Alone and With Exercise Training on Skeletal Muscle Function in the Elderly
Brief Title: Clinical Trial of Astaxanthin Formulation With Exercise in Sarcopenia Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Astavita, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ax sarcopenia study
Record Dates: First submitted 2017-12-06; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Sarcopenia
Keywords: Sarcopenia, muscle function, muscle endurance, fatigue
MeSH Terms: conditions — Sarcopenia; Fatigue | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astaxanthin and exercise (Experimental): Astaxanthin formulation intake for one month followed by a 3-month exercise training program with astaxanthin formulation intake.
  Interventions: Other: Astaxanthin formulation; Other: Exercise training
- Placebo and exercise (Placebo Comparator): Placebo intake for one month followed by 3-month exercise training with placebo intake.
  Interventions: Other: Placebo; Other: Exercise training

INTERVENTIONS:
Other: Astaxanthin formulation — Astaxanthin formulation containing AstaReal® astaxanthin (Haematococcus pluvialis algae extract), tocotrienol, and zinc will be orally administered starting on Day 1 until Day 120
  Other Names: AstaMed MYO
  Arms: Astaxanthin and exercise
Other: Placebo — Placebo will be orally administered starting on Day 1 until Day 120.
  Arms: Placebo and exercise
Other: Exercise training — The subjects will undergo interval treadmill incline protocol (target 85% HR max, 3 times a week for 40 to 60 minutes) starting on Day 31 until Day 120.

SUMMARY:
The primary objective of this trial is to evaluate the effect of oral administration of an Astaxanthin formulation compared to placebo after one month alone and after an additional 3 months of exercise training on mitochondrial and skeletal muscle function in elderly subjects with evidence of mitochondrial dysfunction/sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Able to travel to and from the study facilities
* Informed consent obtained

Exclusion Criteria:

* Have significant disease(s) or condition(s) which, in the opinion of the investigator, may put the subject at risk because of their participation in the trial or may influence either the results of the trial or the subject's ability to participate in the trial
* Hospitalization within 3 months for major atherosclerotic events (defined as combined incidence of myocardial infarction, urgent target-vessel revascularization, coronary bypass surgery and stroke) and for any hospitalization within 2 months.
* Have any metal implant in the right upper limb, including metal stents, titanium pins/markers, etc.
* Have an implanted cardiac pacemaker or other implanted cardiac device
* Chronic, uncontrolled hypertension as judged by the Investigator (ie, Baseline SBP >150 mm Hg, DBP >90 mm Hg) or a SBP > 150 mm Hg or DBP > 95 mm Hg at the time of screening or baseline. If the initial BP reading is above these values, the reading may be repeated one time within 20 minutes of the initial reading.
* Body mass index <18 or >32 kg/m2
* Creatinine clearance calculated by the Cr/G method calculated to be <45 mL/min
* Additional laboratory abnormalities determined as clinically significant by the Investigator Clinically significant abnormalities on physical examination (as judged by the Investigator)
* History or evidence of renal, hepatic, pulmonary (including chronic asthma), endocrine (eg, diabetes, hypo- and hyperthyroidism, adrenal insufficiency), central nervous or neurologic disorders (MS, epilepsy, history of seisures), or gastrointestinal (cirrhosis or viral hepatitis) system dysfunction
* History of seizures or epilepsy
* History of serious mental illness as judged by the Investigator
* Oral temperature >37.5°C at the time of the physical
* Suspicion, or recent history, of alcohol or substance abuse or tobacco use, including positive results from the laboratory screening panels conducted at screening
* Donated blood or blood products within the past 30 days
* Subjects who in the opinion of the Investigator have a clinically significant abnormal 12-lead ECG during the screening period. Presence of atrial fibrillation, varying degrees of AV block, existence of a left bundle branch block, or evidence of previous myocardial infarction.
* Subjects who are either unwilling to agree to refrain from using or found to be using supplementary antioxidant vitamins (eg, Coenzyme Q10) from 7 days prior to dosing and throughout the confinement period
* Are currently enrolled in a clinical trial involving an investigational product or non approved use of a drug or device or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study Have participated, within the last 30 days from a clinical trial involving an investigational product. If the previous investigational product has a long half life, 3 months or 5 half-lives (whichever is longer) should have passed

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle strength and performance measured by 31P-magnetic resonance spectroscopy (31p MRS) | Day 30 - Day 120
  Skeletal muscle strength and performance will be evaluated by changes from baseline in muscle work rate calculated from the results of the leg muscle fatigue protocol testing: Baseline-Day 30-Day 120.

SECONDARY OUTCOMES:
Muscle energetics | Day 30-Day 120
  Muscle energetics and size measured by 31p MRS: Baseline
Hand grip strength | Day 30-Day120
  Hand grip strength
6-minute walk test | Day 30-Day 120
  6-minute walk test
Safety Measures | Baseline-Day 30-Day 120
  Safety as assessed by measures such as adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center Prevention Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No